CLINICAL TRIAL: NCT01229540
Title: Clinical Research on Retinal Neovascularization of Diabetic Retinopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University (Other)
Other Study IDs: 08ZCGYSF01700; 08ZCGYSF01700 (Other: Tianjin Science and Technology Commission)
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2008-09

CONDITIONS: The Mechanism of Retinal Neovascularization of Diabetic; Retinopathy.
MeSH Terms: conditions — Retinal Diseases

ARMS (1):
- Lifestyle counseling (No Intervention)
  Interventions: Genetic: genetic analyzer

INTERVENTIONS:
Genetic: genetic analyzer

SUMMARY:
Retinal neovascularization of diabetic retinopathy might be associated with genetic risk factors and environmental risk factors.

ELIGIBILITY:
Inclusion Criteria:

* T2DM was diagnosed according to the World Health Organization Expert Consultation Report 1999 and consisted of one of the following: fasting blood glucose (FBG) ≥7.0 mmol/L (≥126 mg/dL), blood glucose ≥11.1 mmol/L (≥200 mg/dL) 2 hours after an oral glucose tolerance test (OGTT); or a random blood glucose ≥11.1 mmol/L (≥200 mg/dL).
* DR was clinically graded in accordance with the International Clinical Diabetic Retinopathy guidelines based on fundus fluorescence angiography.
* All participants with PDR underwent a comprehensive dilated fundus examination to detect DR by indirect ophthalmoscopy and were diagnosed by fundus fluorescence angiography.

Exclusion Criteria:

* Patients were excluded if they had acute complications of diabetes mellitus, type 1 diabetes mellitus, other types of diabetes, serious cardiovascular, hepatic, nephritic or other complications, other serious primary diseases or mental illness.

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Clinical college of Ophthalmology ,Tianjin Medical Univercity, Tianjin, Tianjin Municipality, China